CLINICAL TRIAL: NCT01193413
Title: Soluble Triggering Receptor Expressed on Myeloid Cells in Severe Acute Pancreatitis: a Marker of Infected Necrosis and Indicator of Treatment
Brief Title: Soluble Triggering Receptor Expressed on Myeloid Cells in Severe Acute Pancreatitis
Acronym: STREM-1
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Zhaoshen Li, Changhai Hospital, Second Military Medical University
Other Study IDs: Changhai-100829; 30772138 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2010-08-30; First posted 2010-09-02 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Acute; Pancreatitis
Keywords: acute pancreatitis; Drainage; Pancreatic surgery; Biological Markers/analysis; Infection diagnosis; ROC Curve; Sensitivity and Specificity; Endoscopic ultrasonography
MeSH Terms: conditions — Pancreatitis; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The FNA fluid specimens were performed under ultrasound or CT guidance, using a 18G needle attached to a 15 ml eppendorf tube. One percent xylocaine was used for local anaesthesia. Under real-time visualization, the needle was directed into the tissue part of the necrosis or pseudocyst.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Non-infected necrosis group: There is no necrosis infection in severe acute pancreatitis.
- Single drainage group: The patients with necrosis infection in severe acue pancreatitis were cured by single drainage.
- Combined surgery group: If there was no clinical improvement after single drainage about 7 days, an open necrosectomy was performed in the patients with necrosis infection.

SUMMARY:
Early diagnosis of secondary infection of necrotic tissue in severe acute pancreatitis is extremely important. The investigators evaluated whether the level of soluble TREM-1 (sTREM-1) in fine needle aspiration (FNA) fluid from patients who suspected infection is a good marker of secondary infection of necrotic tissue and an indicator of the proper treatment between drainage and necrosectomy.

DETAILED DESCRIPTION:
The major cause of death, next to early organ failure, is secondary infection of pancreatic or peripancreatic necrotic tissue, leading to sepsis and multiple organ failure. The diagnosis and treatment of infected necrosis in SAP remain a major challenge for clinicians. The necrotic infection is defined when microorganisms are isolated from the samples of ultrasound or computed tomography (CT) guided fine needle aspiration (FNA). Unfortunately, a negative biopsy result can not completely rule out infection and the repeated aspirations may lead to bleeding or iatrogenic infection. Moreover, whatever the microbiologic diagnostic procedure chosen, further laboratory processing and delays of 24 to 48 hours are required for definitive quantitative microbial culture results. Meanwhile, clinicians often feel uncomfortable about the diagnosis and may administer unneeded antibiotics while awaiting laboratory results.

Secondary infection of necrotic tissue in SAP patients is virtually always an indication for intervention. The traditional approach is open necrosectomy to completely remove the infected necrotic tissue. This invasive approach is associated with high rates of complications (34 to 95%) and death (11 to 39%).As an alternative to open necrosectomy, less invasive techniques, including percutaneous drainage and endoscopic (transgastric) drainage, are increasingly being used.These steps may postpone or even obviate surgical necrosectomy with reducing complications and death.It remains uncertain which intervention is optimal in terms of clinical conditions of these patients and the severity of local infection.

Therefore, many biologic markers have been studied in an effort to improve the diagnostic rate and determine the the severity of necrosis infection but with disappointing results. The triggering receptor expressed on myeloid cells (TREM-1) is a member of the immunoglobulin superfamily whose expression on phagocytes is up-regulated by exposure to bacteria and fungi. TREM-1 mediates the acute inflammatory response to microbial products.[27] TREM-1 is also shed by the membrane of activated phagocytes and can be found in a soluble form in body fluids. We evaluated whether the lever of soluble TREM-1 (sTREM-1) in FNA fluid from patients who suspected infection is a good marker of secondary infection of necrotic tissue and an indicator of the proper treatment between drainage and necrosectomy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of severe pancreatitis
* Pancreatic or peripancreatic necrosis
* Body temperature at least 38.3°C
* Leukocytosis (more than 10,000 leukocytes per cubic millimeter) or leukopenia (fewer than 4000 leukocytes per cubic millimeter)

Exclusion Criteria:

* A flare-up of chronic pancreatitis
* End-stage chronic diseases (including pancreatic and bile duct cancer)
* Previous drainage or surgery for confirmed or suspected infected necrosis
* An acute intraabdominal event (e.g., perforation of a visceral organ, bleeding, or the abdominal compartment syndrome)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 18 years of age or older who were hospitalized in our medical pancreatic intensive care unit (PICU) for least two weeks were enrolled in the study if there was a clinical suspicion of secondary infection of necrotic tissue.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The level of sTREM-1 in fine needle aspiration fluid | more than 14 days after entry
  The fluid level of sTREM-1 was used to diagnose the secondary infection of necrotic tissues in severe acute pancreatitis and select the proper treatment between single drainage and necrosectomy.

SECONDARY OUTCOMES:
The fluid level of Interleukin-6 | more than 14 days after entry
  The fluid level of Interleukin-6 was used to diagnose the secondary infection of necrotic tissues in severe acute pancreatitis and select the proper treatment between single drainage and necrosectomy.
The fluid level of tumor necrosis factor-α | more than 14 days after entry
  The fluid level of tumor necrosis factor-α was used to diagnose the secondary infection of necrotic tissues in severe acute pancreatitis and select the proper treatment between single drainage and necrosectomy.
The serum level of sTREM-1 | more than 14 days after entry
  The serum level of sTREM-1 was used to diagnose the secondary infection of necrotic tissues in severe acute pancreatitis and select the proper treatment between single drainage and necrosectomy.
The serum level of C-reactive protein | more than 14 days after entry
  The serum level of C-reactive protein was used to diagnose the secondary infection of necrotic tissues in severe acute pancreatitis and select the proper treatment between single drainage and necrosectomy.
The level of leukocyte count and neutrophil percentage | more than 14 days after entry
  The level of leukocyte count and neutrophil percentage was used to diagnose the secondary infection of necrotic tissues in severe acute pancreatitis and select the proper treatment between single drainage and necrosectomy.

CONTACTS AND LOCATIONS:
Overall Officials: zhaoshen li, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China